CLINICAL TRIAL: NCT02516280
Title: Effects of Hyperbaric Gaseous Cryotherapy on Knee Flexion Range of Motion in the First Two Days After Total Knee Arthroplasty: A Feasibility Randomized Controlled Trial
Brief Title: Effects of Gaseous Cryotherapy on Knee ROM After TKA: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Verdun (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHV2012-01
Record Dates: First submitted 2015-07-27; First posted 2015-08-05 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Osteoarthritis, Knee
Keywords: Total knee replacement; Cold; Neurocryostimulation; CO2 cryotherapy; mobility
MeSH Terms: conditions — Osteoarthritis, Knee; Common Cold | interventions — Cryopreservation; Dental Pulp Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyperbaric gaseous cryotherapy group (Experimental): Conventional rehabilitation with Cryoton ™ hyperbaric cryotherapy
  Interventions: Device: Cryoton ™
- Control ice bag group (Active Comparator): Conventional rehabilitation with ice bag cryotherapy. Application of a bag of crushed ice directly on the anterior aspect of the knee.
  Interventions: Device: Control ice bag

INTERVENTIONS:
Device: Cryoton ™ — In the intervention group, participants received hyperbaric gaseous cryotherapy delivered with a Cryoton ™ device (Cryonic Médical, Salins-les-Bains, France) within an hour after the surgery and two times per day the next postoperative days. The tip of the nozzle was kept 10-15 cm above the dry skin as the gaseous CO2 was sprayed on three zones of 5 cm by 10 cm (medial, lateral and posterior, respectively) using a slow and regular sweeping movement for approximately 30 seconds after a skin temperature of 2°C is reached.
  Other Names: Neurocryostimulation; Cryonic
  Arms: Hyperbaric gaseous cryotherapy group
Device: Control ice bag — In the control group, participants received two 20-minute treatments of cryotherapy within an hour after the surgery and two times per day the next postoperative days. Cryotherapy was performed using an ice bag that was applied directly on the anterior aspect of the knee. The ice bag is a square latex bag of 30 cm by 30 cm filled with crushed ice and wrapped in a thin pillow case. The treatment assessor applied the intervention in a standardized manner by ensuring that the knee was fully extended while covering the surgical incision and both lateral and medial aspects of the knee with the iced bag.
  Other Names: ice
  Arms: Control ice bag group

SUMMARY:
A pilot study was performed to investigate the feasibility of a large randomized controlled trial (RCT) to assess the effects of hyperbaric gaseous cryotherapy (HGC) on the change in knee flexion range of motion in the first two days after total knee arthroplasty.

DETAILED DESCRIPTION:
Background: After total knee arthroplasty (TKA), patients can be discharged from hospital as early as two days after surgery. However, patients often do not achieve functional knee flexion range of motion (ROM) in the first postoperative days. Early application of hyperbaric gaseous cryotherapy (HGC) at the operated knee within an hour after surgery and the next postoperative days might increase ROM by reducing inflammation, edema and pain. However, it is unclear whether such early application of HGC is feasible. Moreover, there is no data to allow calculation of the sample size required to conduct a randomized controlled trial to compare the effects of HGC to those of conventional cryotherapy on the increase of knee flexion in the first two days after TKA.

Objectives: To investigate the feasibility of applying HGC within an hour after TKA and twice a day the next postoperative days. To collect data on changes in knee flexion ROM in the first two postoperative days to calculate the sample size required for a large randomized controlled trial. To compare the effects of HGC to those of conventional cryotherapy on changes in knee flexion ROM in the first two postoperative days.

Design: A prospective, single-blinded, randomized, controlled pilot trial.

Setting: Orthopedic postoperative unit in an acute care hospital.

Interventions: Patients were randomly allocated to either hyperbaric gaseous cryotherapy (intervention group) or the ice bag cryotherapy (control group). In each group, participants received the specific cryotherapy intervention at the operated knee within an hour after the surgery (day 0) and twice the next two postoperative days (day 1 and day 2).

Outcome measures: Feasibility measures included the rate of eligible patients who were willing to participate, attrition, adherence to interventions and presence of adverse effects. Active and passive knee flexion range of motion (ROM) and knee pain intensity at rest were evaluated on postoperative days 1 and 2. Change in active and passive knee flexion ROM and in knee pain intensity at rest from postoperative day 1 to day 2 were assessed. Length of hospital stay was collected.

ELIGIBILITY:
Inclusion Criteria:

* Planned unilateral TKA done at Verdun Hospital.
* Capacity to communicate in French or English.

Exclusion Criteria:

* Complications during or after the surgery.
* Inability to perform the tests due to other diseases.
* Contraindications to cryotherapy such as Raynaud's disease, cryoglobulinemia, hemoglobinopathy, polyneuropathy associated with temperature sensitivity deficits or allergy to cold.

Ages: 35 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Changes in active and passive knee flexion ROM measured by analysis. | Between post-operative day 1 and 2
  The primary outcomes were changes in active and passive knee flexion ROM from postoperative day 1 to day 2. This outcome was calculated as the difference in active and passive ROM between day 2 and day 1

SECONDARY OUTCOMES:
Active and passive knee flexion ROM measured using goniometry. | During the first 2 days after surgery.
  Active and passive knee flexion ROMs were measured with a long-arm (35 cm) goniometer featuring a 360º and two 180º scales, with 1º increments that read in opposite directions (Baseline 360° 14" Goniometer, Fabrication enterprises Inc., NY, USA). Knee ROMs were measured in sitting position because levels of agreement between observers are higher in sitting position than in supine position.
Knee pain measured by visual analog scale. | During the first 2 days after surgery.
  Scale from 0 to 10 cm on a ruler where 0 represented no pain and 10 represented the worst pain imaginable.
Change in pain from postoperative day 1 to day 2 measured by analysis of variation of the recorded pain between data of day2 and day 1 (Knee pain measured by visual analog scale) | Between day 1 and 2.
  Calculated as the difference of pain between day 2 and day 1.
Feasibility was assessed by analysis of presence of adverse effects. | Participants will be followed for the duration of hospital stay, an expected average of 3 days.
  Determine if the patients where having or not adverse during thier stay.
Feasibility was assessed by adherence to the intervention (attrition). | Participants will be followed for the duration of hospital stay, an expected average of 3 days.
  Determine if the patients where adhering to treatment (drop-off).
Length of the stay in hospital ward was measured by the length(in days) of inpatient episode of care. | Participants will be followed for the duration of hospital stay, an expected average of 3 days.
  Length of stay in hospital ward.

CONTACTS AND LOCATIONS:
Overall Officials: David Moreau, MSc, Principal Investigator — Centre Hospitalier de Verdun

REFERENCES:
- [Background] Abramson DI, Chu LS, Tuck S Jr, Lee SW, Richardson G, Levin M. Effect of tissue temperatures and blood flow on motor nerve conduction velocity. JAMA. 1966 Dec 5;198(10):1082-8. No abstract available. PMID 5953385
- [Background] Adie S, Kwan A, Naylor JM, Harris IA, Mittal R. Cryotherapy following total knee replacement. Cochrane Database Syst Rev. 2012 Sep 12;(9):CD007911. doi: 10.1002/14651858.CD007911.pub2. PMID 22972114
- [Background] Adie S, Naylor JM, Harris IA. Cryotherapy after total knee arthroplasty a systematic review and meta-analysis of randomized controlled trials. J Arthroplasty. 2010 Aug;25(5):709-15. doi: 10.1016/j.arth.2009.07.010. Epub 2009 Sep 2. PMID 19729279
- [Background] Alcelik I, Sukeik M, Pollock R, Misra A, Shah P, Armstrong P, Dhebar MI. Comparison of the minimally invasive and standard medial parapatellar approaches for primary total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2012 Dec;20(12):2502-12. doi: 10.1007/s00167-012-1944-3. Epub 2012 Mar 15. PMID 22419264
- [Background] Ayalon O, Liu S, Flics S, Cahill J, Juliano K, Cornell CN. A multimodal clinical pathway can reduce length of stay after total knee arthroplasty. HSS J. 2011 Feb;7(1):9-15. doi: 10.1007/s11420-010-9164-1. Epub 2010 May 22. PMID 22294952
- [Background] Bade MJ, Kittelson JM, Kohrt WM, Stevens-Lapsley JE. Predicting functional performance and range of motion outcomes after total knee arthroplasty. Am J Phys Med Rehabil. 2014 Jul;93(7):579-85. doi: 10.1097/PHM.0000000000000065. PMID 24508937
- [Background] Bade MJ, Kohrt WM, Stevens-Lapsley JE. Outcomes before and after total knee arthroplasty compared to healthy adults. J Orthop Sports Phys Ther. 2010 Sep;40(9):559-67. doi: 10.2519/jospt.2010.3317. PMID 20710093
- [Background] Basso DM, Knapp L. Comparison of two continuous passive motion protocols for patients with total knee implants. Phys Ther. 1987 Mar;67(3):360-3. doi: 10.1093/ptj/67.3.360. PMID 3823150
- [Background] Belitsky RB, Odam SJ, Hubley-Kozey C. Evaluation of the effectiveness of wet ice, dry ice, and cryogenic packs in reducing skin temperature. Phys Ther. 1987 Jul;67(7):1080-4. doi: 10.1093/ptj/67.7.1080. PMID 3602101
- [Background] Bonutti PM, Mont MA, Kester MA. Minimally invasive total knee arthroplasty: a 10-feature evolutionary approach. Orthop Clin North Am. 2004 Apr;35(2):217-26. doi: 10.1016/j.ocl.2004.02.001. PMID 15062707
- [Background] Chatap G, De Sousa A, Giraud K, Vincent JP; Acute Pain in the Elderly Study Group. Pain in the elderly: Prospective study of hyperbaric CO2 cryotherapy (neurocryostimulation). Joint Bone Spine. 2007 Dec;74(6):617-21. doi: 10.1016/j.jbspin.2006.10.011. Epub 2007 Jul 19. PMID 17897861
- [Background] Cheng T, Liu T, Zhang G, Peng X, Zhang X. Does minimally invasive surgery improve short-term recovery in total knee arthroplasty? Clin Orthop Relat Res. 2010 Jun;468(6):1635-48. doi: 10.1007/s11999-010-1285-9. Epub 2010 Mar 13. PMID 20229136
- [Background] Chesterton LS, Foster NE, Ross L. Skin temperature response to cryotherapy. Arch Phys Med Rehabil. 2002 Apr;83(4):543-9. doi: 10.1053/apmr.2002.30926. PMID 11932859
- [Background] Chiu KY, Ng TP, Tang WM, Yau WP. Review article: knee flexion after total knee arthroplasty. J Orthop Surg (Hong Kong). 2002 Dec;10(2):194-202. doi: 10.1177/230949900201000215. PMID 12493934
- [Background] Ciolek JJ. Cryotherapy. Review of physiological effects and clinical application. Cleve Clin Q. 1985 Summer;52(2):193-201. doi: 10.3949/ccjm.52.2.193. No abstract available. PMID 3896574
- [Background] Corbett KL, Reichmann WM, Katz JN, Beagan C, Corsello P, Ghazinouri R, Dang B, Mikulinsky R, Losina E, Wright J. One-Day vs Two-Day Epidural Analgesia for Total Knee Arthroplasty (TKA): A Retrospective Cohort Study. Open Orthop J. 2010 Jan 19;4:31-8. doi: 10.2174/1874325001004010031. PMID 20361034
- [Background] Dayton MR, Bade MJ, Muratore T, Shulman BC, Kohrt WM, Stevens-Lapsley JE. Minimally invasive total knee arthroplasty: surgical implications for recovery. J Knee Surg. 2013 Jun;26(3):195-201. doi: 10.1055/s-0032-1327449. Epub 2012 Nov 12. PMID 23288738
- [Background] Demoulin C, Brouwers M, Darot S, Gillet P, Crielaard JM, Vanderthommen M. Comparison of gaseous cryotherapy with more traditional forms of cryotherapy following total knee arthroplasty. Ann Phys Rehabil Med. 2012 May;55(4):229-40. doi: 10.1016/j.rehab.2012.03.004. Epub 2012 Apr 5. English, French. PMID 22516265
- [Background] Ekenvall L, Lindblad LE, Norbeck O, Etzell BM. alpha-Adrenoceptors and cold-induced vasoconstriction in human finger skin. Am J Physiol. 1988 Nov;255(5 Pt 2):H1000-3. doi: 10.1152/ajpheart.1988.255.5.H1000. PMID 2903677
- [Background] Ernst E, Fialka V. Ice freezes pain? A review of the clinical effectiveness of analgesic cold therapy. J Pain Symptom Manage. 1994 Jan;9(1):56-9. doi: 10.1016/0885-3924(94)90150-3. PMID 8169463
- [Background] Fatoye FA, Palmer ST, Macmillan F, Rowe PJ, van der Linden ML. Repeatability of joint proprioception and muscle torque assessment in healthy children and in children diagnosed with hypermobility syndrome. Musculoskeletal Care. 2008 Jun;6(2):108-23. doi: 10.1002/msc.127. PMID 18348137
- [Background] Freedman RR, Sabharwal SC, Moten M, Migaly P. Local temperature modulates alpha 1- and alpha 2-adrenergic vasoconstriction in men. Am J Physiol. 1992 Oct;263(4 Pt 2):H1197-200. doi: 10.1152/ajpheart.1992.263.4.H1197. PMID 1329562
- [Background] Garstang SV, Stitik TP. Osteoarthritis: epidemiology, risk factors, and pathophysiology. Am J Phys Med Rehabil. 2006 Nov;85(11 Suppl):S2-11; quiz S12-4. doi: 10.1097/01.phm.0000245568.69434.1a. No abstract available. PMID 17079976
- [Background] Harris ED Jr, McCroskery PA. The influence of temperature and fibril stability on degradation of cartilage collagen by rheumatoid synovial collagenase. N Engl J Med. 1974 Jan 3;290(1):1-6. doi: 10.1056/NEJM197401032900101. No abstract available. PMID 4357162
- [Background] Ho SS, Coel MN, Kagawa R, Richardson AB. The effects of ice on blood flow and bone metabolism in knees. Am J Sports Med. 1994 Jul-Aug;22(4):537-40. doi: 10.1177/036354659402200417. PMID 7943521
- [Background] Husted H, Holm G, Jacobsen S. Predictors of length of stay and patient satisfaction after hip and knee replacement surgery: fast-track experience in 712 patients. Acta Orthop. 2008 Apr;79(2):168-73. doi: 10.1080/17453670710014941. PMID 18484241
- [Background] Insall J. A midline approach to the knee. J Bone Joint Surg Am. 1971 Dec;53(8):1584-6. No abstract available. PMID 5121799
- [Background] Kennedy DM, Stratford PW, Wessel J, Gollish JD, Penney D. Assessing stability and change of four performance measures: a longitudinal study evaluating outcome following total hip and knee arthroplasty. BMC Musculoskelet Disord. 2005 Jan 28;6:3. doi: 10.1186/1471-2474-6-3. PMID 15679884
- [Background] Kettelkamp DB, Johnson RJ, Smidt GL, Chao EY, Walker M. An electrogoniometric study of knee motion in normal gait. J Bone Joint Surg Am. 1970 Jun;52(4):775-90. No abstract available. PMID 5479460
- [Background] Kim J, Seo BS. How to calculate sample size and why. Clin Orthop Surg. 2013 Sep;5(3):235-42. doi: 10.4055/cios.2013.5.3.235. Epub 2013 Aug 20. PMID 24009911
- [Background] Knight KL, Londeree BR. Comparison of blood flow in the ankle of uninjured subjects during therapeutic applications of heat, cold, and exercise. Med Sci Sports Exerc. 1980 Spring;12(1):76-80. doi: 10.1249/00005768-198021000-00015. PMID 6771484
- [Background] Kurtz SM, Ong KL, Lau E, Widmer M, Maravic M, Gomez-Barrena E, de Pina Mde F, Manno V, Torre M, Walter WL, de Steiger R, Geesink RG, Peltola M, Roder C. International survey of primary and revision total knee replacement. Int Orthop. 2011 Dec;35(12):1783-9. doi: 10.1007/s00264-011-1235-5. Epub 2011 Mar 15. PMID 21404023
- [Background] Laubenthal KN, Smidt GL, Kettelkamp DB. A quantitative analysis of knee motion during activities of daily living. Phys Ther. 1972 Jan;52(1):34-43. doi: 10.1093/ptj/52.1.34. No abstract available. PMID 5061683
- [Background] Lenssen AF, Crijns YH, Waltje EM, van Steyn MJ, Geesink RJ, van den Brandt PA, de Bie RA. Efficiency of immediate postoperative inpatient physical therapy following total knee arthroplasty: an RCT. BMC Musculoskelet Disord. 2006 Aug 31;7:71. doi: 10.1186/1471-2474-7-71. PMID 16942627
- [Background] Lenssen AF, van Dam EM, Crijns YH, Verhey M, Geesink RJ, van den Brandt PA, de Bie RA. Reproducibility of goniometric measurement of the knee in the in-hospital phase following total knee arthroplasty. BMC Musculoskelet Disord. 2007 Aug 17;8:83. doi: 10.1186/1471-2474-8-83. PMID 17705860
- [Background] Lin YC, Davey RC, Cochrane T. Tests for physical function of the elderly with knee and hip osteoarthritis. Scand J Med Sci Sports. 2001 Oct;11(5):280-6. doi: 10.1034/j.1600-0838.2001.110505.x. PMID 11696212
- [Background] Markert SE. The use of cryotherapy after a total knee replacement: a literature review. Orthop Nurs. 2011 Jan-Feb;30(1):29-36. doi: 10.1097/NOR.0b013e318205749a. PMID 21278552
- [Background] Martin SS, Spindler KP, Tarter JW, Detwiler KB. Does cryotherapy affect intraarticular temperature after knee arthroscopy? Clin Orthop Relat Res. 2002 Jul;(400):184-9. doi: 10.1097/00003086-200207000-00023. PMID 12072761
- [Background] McKay C, Prapavessis H, Doherty T. The effect of a prehabilitation exercise program on quadriceps strength for patients undergoing total knee arthroplasty: a randomized controlled pilot study. PM R. 2012 Sep;4(9):647-56. doi: 10.1016/j.pmrj.2012.04.012. Epub 2012 Jun 13. PMID 22698852
- [Background] McLean DA. The use of cold and superficial heat in the treatment of soft tissue injuries. Br J Sports Med. 1989 Mar;23(1):53-4. doi: 10.1136/bjsm.23.1.53. No abstract available. PMID 2731001
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Mizner RL, Petterson SC, Stevens JE, Vandenborne K, Snyder-Mackler L. Early quadriceps strength loss after total knee arthroplasty. The contributions of muscle atrophy and failure of voluntary muscle activation. J Bone Joint Surg Am. 2005 May;87(5):1047-53. doi: 10.2106/JBJS.D.01992. PMID 15866968
- [Background] Mourot L, Cluzeau C, Regnard J. Hyperbaric gaseous cryotherapy: effects on skin temperature and systemic vasoconstriction. Arch Phys Med Rehabil. 2007 Oct;88(10):1339-43. doi: 10.1016/j.apmr.2007.06.771. PMID 17908579
- [Background] Mourot L, Cluzeau C, Regnard J. [Physiological assessment of a gaseous cryotherapy device: thermal effects and changes in cardiovascular autonomic control]. Ann Readapt Med Phys. 2007 May;50(4):209-17. doi: 10.1016/j.annrmp.2007.01.005. Epub 2007 Jan 26. French. PMID 17300850
- [Background] Nutton RW, Wade FA, Coutts FJ, van der Linden ML. Short Term Recovery of Function following Total Knee Arthroplasty: A Randomised Study of the Medial Parapatellar and Midvastus Approaches. Arthritis. 2014;2014:173857. doi: 10.1155/2014/173857. Epub 2014 Oct 1. PMID 25349736
- [Background] Ohkoshi Y, Ohkoshi M, Nagasaki S, Ono A, Hashimoto T, Yamane S. The effect of cryotherapy on intraarticular temperature and postoperative care after anterior cruciate ligament reconstruction. Am J Sports Med. 1999 May-Jun;27(3):357-62. doi: 10.1177/03635465990270031601. PMID 10352774
- [Background] Oldmeadow LB, McBurney H, Robertson VJ. Hospital stay and discharge outcomes after knee arthroplasty: implications for physiotherapy practice. Aust J Physiother. 2002;48(2):117-21. doi: 10.1016/s0004-9514(14)60205-1. PMID 12047209
- [Background] Olson JE, Stravino VD. A review of cryotherapy. Phys Ther. 1972 Aug;52(8):840-53. doi: 10.1093/ptj/52.8.840. No abstract available. PMID 4558889
- [Background] Pavlov VA, Tracey KJ. The cholinergic anti-inflammatory pathway. Brain Behav Immun. 2005 Nov;19(6):493-9. doi: 10.1016/j.bbi.2005.03.015. PMID 15922555
- [Background] Raynor MC, Pietrobon R, Guller U, Higgins LD. Cryotherapy after ACL reconstruction: a meta-analysis. J Knee Surg. 2005 Apr;18(2):123-9. doi: 10.1055/s-0030-1248169. PMID 15915833
- [Background] Remy C, Marret E, Bonnet F. Effects of acetaminophen on morphine side-effects and consumption after major surgery: meta-analysis of randomized controlled trials. Br J Anaesth. 2005 Apr;94(4):505-13. doi: 10.1093/bja/aei085. Epub 2005 Jan 28. PMID 15681586
- [Background] Salinas FV, Liu SS, Mulroy MF. The effect of single-injection femoral nerve block versus continuous femoral nerve block after total knee arthroplasty on hospital length of stay and long-term functional recovery within an established clinical pathway. Anesth Analg. 2006 Apr;102(4):1234-9. doi: 10.1213/01.ane.0000198675.20279.81. PMID 16551930
- [Background] Scarcella JB, Cohn BT. The effect of cold therapy on the postoperative course of total hip and knee arthroplasty patients. Am J Orthop (Belle Mead NJ). 1995 Nov;24(11):847-52. PMID 8581442
- [Background] Singelyn FJ, Ferrant T, Malisse MF, Joris D. Effects of intravenous patient-controlled analgesia with morphine, continuous epidural analgesia, and continuous femoral nerve sheath block on rehabilitation after unilateral total-hip arthroplasty. Reg Anesth Pain Med. 2005 Sep-Oct;30(5):452-7. doi: 10.1016/j.rapm.2005.05.008. PMID 16135349
- [Background] Stevens-Lapsley JE, Balter JE, Wolfe P, Eckhoff DG, Kohrt WM. Early neuromuscular electrical stimulation to improve quadriceps muscle strength after total knee arthroplasty: a randomized controlled trial. Phys Ther. 2012 Feb;92(2):210-26. doi: 10.2522/ptj.20110124. Epub 2011 Nov 17. PMID 22095207
- [Background] Thorsson O, Lilja B, Ahlgren L, Hemdal B, Westlin N. The effect of local cold application on intramuscular blood flow at rest and after running. Med Sci Sports Exerc. 1985 Dec;17(6):710-3. doi: 10.1249/00005768-198512000-00016. PMID 4079745
- [Background] Webb JM, Williams D, Ivory JP, Day S, Williamson DM. The use of cold compression dressings after total knee replacement: a randomized controlled trial. Orthopedics. 1998 Jan;21(1):59-61. doi: 10.3928/0147-7447-19980101-14. PMID 9474633
- [Background] Zachariassen KE. Hypothermia and cellular physiology. Arctic Med Res. 1991;50 Suppl 6:13-7. PMID 1811567